CLINICAL TRIAL: NCT02715700
Title: A Multiple-Dose Clinical Trial to Study the Effect of MK-1439 (Doravirine) on Methadone Pharmacokinetics
Brief Title: Effects of Doravirine (MK-1439) on Methadone Pharmacokinetics in Methadone-Maintained Participants (MK-1439-045)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1439-045; MK-1439-045 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Methadone; doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maintenance Methadone and MK-1439 (Experimental): Participants maintained on a stable methadone regimen (20 to 200 mg once daily) for ≥14 days prior to Day 1 will continue to receive methadone maintenance once per day on Days 1 to 7. From Day 2 to 6, participants will also receive doravirine 100 mg once daily.
  Interventions: Drug: Methadone; Drug: Doravirine

INTERVENTIONS:
Drug: Methadone — Methadone 20 to 200 mg (10 mg/mL if oral solution concentrate) oral tablet once per day.
Drug: Doravirine — Doravirine 100 mg oral tablet once per day.
  Other Names: MK-1439

SUMMARY:
This study will evaluate the effects of multiple doses of doravirine (MK-1439) on the pharmacokinetics of methadone in participants requiring methadone maintenance therapy. The primary hypothesis is that area under the plasma concentration-time curve to 24 hours postdose (AUC0-24) of (R)-methadone is similar when a maintenance regimen of methadone is administered with or without multiple daily doses of doravirine.

ELIGIBILITY:
Inclusion Criteria:

* If female with reproductive potential: must demonstrate a serum β-human chorionic gonadotropin (β -hCG) level consistent with the nongravid state and agree to use (and/or have their partner use) two acceptable methods of birth control throughout the trial and until 2 weeks after the last dose of trial drug.
* If postmenopausal female: must be without menses for at least 1 year.
* If surgically sterile female: must have a status of post hysterectomy, oophorectomy or tubal ligation.
* Body Mass Index (BMI) of 18-35 kg/m^2 (inclusive).
* Able to comply with the smoking restrictions, including <=10 cigarettes per day while in the Clinical Research Unit, and no smoking from 2 hours predose to 2 hours postdose on Days 1 and 6.
* Reliably participating in a methadone maintenance program for at least two months prior to Day 1. Required to be on a documented stable dose of methadone for at least 14 days prior to Day 1.
* Agree not to change current maintenance methadone dose of 20-200 mg once daily (unless for safety reasons) from screening until the end of the study. Must agree to observation and documentation of daily methadone dose administration during the period of the study during which they are domiciled.

Exclusion Criteria:

* Mentally or legally incapacitated, have significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or have a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the trial at the discretion of the investigator.
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a history of uncomplicated kidney stones or childhood asthma may be enrolled in the trial at the discretion of the investigator.
* History of cancer (malignancy) - exceptions apply.
* History of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Positive for Human Immunodeficiency Virus (HIV).
* Major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* Participated in another investigational trial within 4 weeks prior to the pretrial (screening) visit.
* Nursing mother.
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to the first dose of the 14 day methadone maintenance phase prior to Day 1, throughout the trial, until the post-trial visit - exceptions apply.
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day - exceptions apply.
* Consumes excessive amounts of caffeine, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day.
* Has a positive screen for drugs with a high potential for abuse such as cocaine, amphetamines, methylenedioxymethamphetamine (MDMA), barbiturates, benzodiazepines (exceptions apply), or opiates/opioids (apart from methadone as assigned maintenance therapy) on Day 1 that cannot be explained by concomitant medications, unless at the discretion of the principal investigator and the sponsor. Must have a negative Urine Drug Screen prior to randomization, with the exception of tetrahydrocannabinol (THC) and prescription benzodiazepines.
* Clinical Opiate Withdrawal Scale (COWS) score of >=5 prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Khalilieh S, Yee KL, Sanchez RI, Vaynshteyn K, Fan L, Searle S, Bouhajib M, Iwamoto M. Evaluation of the Pharmacokinetic Interaction Between Doravirine and Methadone. Clin Pharmacol Drug Dev. 2020 Feb;9(2):151-161. doi: 10.1002/cpdd.699. Epub 2019 May 23. PMID 31120195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants on stable methadone maintenance therapy were recruited at 2 study sites in the United States.
Groups:
- Maintenance Methadone + Doravirine: Participants maintained on a stable methadone regimen (20 to 200 mg once daily) for ≥14 days prior to Day 1 received the methadone maintenance dose on Days 1 to 7 and doravirine 100 mg on Days 2 to 6.
Period: Overall Study
Arm/Group | Maintenance Methadone + Doravirine
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Zero to 24 Hours After Dosing (AUC0-24) of R-Methadone
Description: The AUC0-24 of the R- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by liquid chromatographic-tandem mass spectrometric (LC-MS/MS) detection. The lower limit of quantification (LLoQ) was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL/mg
Groups:
- Maintenance Methadone: Participants maintained on a stable methadone regimen (20 to 200 mg once daily) for ≥14 days prior to Day 1 received the methadone maintenance dose on Day 1.
- Maintenance Methadone + Doravirine: Participants maintained on a stable methadone regimen (20 to 200 mg once daily) for ≥14 days prior to Day 1 received the methadone maintenance dose + doravirine 100 mg once daily on Days 2 to 6.
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng*hr/mL/mg | 55.8 [46.4 to 67.1] | 53.2 [44.6 to 63.5]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — Geometric mean ratio (GMR) of Methadone + Doravirine/Methadone Alone; GMR = 0.95, 90% CI 2-sided [0.90 to 1.01]

2. Primary Outcome: Plasma Concentration at 24 Hours After Dosing (C24) of R-Methadone
Description: The C24 of the R- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 1.91 [1.56 to 2.34] | 1.82 [1.45 to 2.27]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.95, 90% CI 2-sided [0.88 to 1.03]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of R-Methadone
Description: The Cmax of the R- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 3.41 [2.89 to 4.01] | 3.33 [2.83 to 3.91]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.98, 90% CI 2-sided [0.93 to 1.03]

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of R-Methadone
Description: The Tmax of the R- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Median (Full Range); unit: Hours
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
Hours | 2.00 [1.00 to 6.00] | 2.01 [1.02 to 4.00]

5. Primary Outcome: AUC0-24 of S-Methadone
Description: The AUC0-24 of the S- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng*hr/mL/mg | 52.0 [38.3 to 70.4] | 50.8 [37.5 to 68.8]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — Geometric mean ratio (GMR) of Methadone + Doravirine/Methadone Alone; GMR = 0.98, 90% CI 2-sided [0.90 to 1.06]

6. Primary Outcome: C24 of S-Methadone
Description: The C24 of the S- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 1.51 [1.03 to 2.22] | 1.47 [0.974 to 2.21]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.97, 90% CI 2-sided [0.86 to 1.10]

7. Primary Outcome: Cmax of S-Methadone
Description: The Cmax of the S- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 3.77 [2.95 to 4.82] | 3.67 [2.87 to 4.68]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.97, 90% CI 2-sided [0.91 to 1.04]

8. Primary Outcome: Tmax of S-Methadone
Description: The Tmax of the S- methadone enantiomer was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Median (Full Range); unit: Hours
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
Hours | 1.99 [1.00 to 3.00] | 2.00 [1.02 to 4.00]

9. Primary Outcome: AUC0-24 of Total Methadone
Description: The AUC0-24 of total methadone was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng*hr/mL/mg | 109 [86.0 to 137] | 105 [82.9 to 132]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — Geometric mean ratio (GMR) of Methadone + Doravirine/Methadone Alone; GMR = 0.96, 90% CI 2-sided [0.90 to 1.03]

10. Primary Outcome: C24 of Total Methadone
Description: The C24 of total methadone was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 3.48 [2.65 to 4.57] | 3.34 [2.48 to 4.51]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.96, 90% CI 2-sided [0.87 to 1.05]

11. Primary Outcome: Cmax of Total Methadone
Description: The Cmax of total methadone was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
ng/mL/mg | 7.19 [5.86 to 8.82] | 7.01 [5.72 to 8.60]
Statistical Analysis 1: Comparison: Maintenance Methadone vs Maintenance Methadone + Doravirine; Test type: Other — GMR of Methadone + Doravirine/Methadone Alone; GMR = 0.98, 90% CI 2-sided [0.92 to 1.03]

12. Primary Outcome: Tmax of Total Methadone
Description: The Tmax of total methadone was determined on Day 1 (methadone alone) and on Day 6 (methadone + doravirine). Plasma samples collected for methadone assay were analyzed for R- and S-methadone concentrations by Pharma Medica Research Inc. (Ontario, Canada). The analytical method used liquid-liquid extraction for analyte isolation followed by LC-MS/MS detection. The LLoQ was 0.0250 ng/mL for each enantiomer. The analytical range was 0.0250 - 15.0 ng/mL.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose on Day 1 and Day 6
Population: All treated participants are included.
Measure: Median (Full Range); unit: Hours
Arm/Group | Maintenance Methadone | Maintenance Methadone + Doravirine
Number analyzed (Participants) | 14 | 14
Hours | 2.00 [1.00 to 6.00] | 2.01 [1.02 to 4.00]

ADVERSE EVENTS:
Time Frame: Up to 21 days
Description: All treated participants are included.
Groups:
- Maintenance Methadone (Day 1): Participants received the methadone maintenance dose on Day 1.
- Maintenance Methadone + Doravirine (Days 2 to 6): Participants received the methadone maintenance dose and doravirine 100 mg on Days 2 to 6.
- Maintenance Methadone (Day 7): Participants received the maintenance methadone dose on Day 7.
- Safety Follow-Up (Days 8 to 21): Participants were monitored for safety for 14 days after the final dose of study treatment.
Arm/Group | Maintenance Methadone (Day 1) | Maintenance Methadone + Doravirine (Days 2 to 6) | Maintenance Methadone (Day 7) | Safety Follow-Up (Days 8 to 21)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 7/14 | 2/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Methadone (Day 1) (N=14) | Maintenance Methadone + Doravirine (Days 2 to 6) (N=14) | Maintenance Methadone (Day 7) (N=14) | Safety Follow-Up (Days 8 to 21) (N=14)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.